CLINICAL TRIAL: NCT05139459
Title: Sepsis in Sub-Saharan Africa: a Prospective Observational Study of Clinical Characteristics, Management, Outcomes, and Barriers to Care in Northern Tanzania
Brief Title: Sepsis Characterization in Kilimanjaro
Acronym: SICK
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00101917; R01AI155733 (NIH)
Record Dates: First submitted 2021-11-11; First posted 2021-12-01 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Sepsis
Keywords: Africa; Tanzania
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be collected in a PaxGene RNA stabilizing tube (BD, Franklin Lakes, New Jersey, USA) at 4 time-points and archived for future studies regarding causes of sepsis or measuring the dysregulated immune response in sepsis, specifically to investigate biomarkers for sepsis mortality and biomarkers to improve triage for sepsis patients in resource-limited settings. These archived samples may also be utilized for etiologic investigations for causes of sepsis using tests for nucleic acid detection or serologic assays.
  Additional specimen archival (at -80 C) will include the following sample types:
  Nasopharyngeal specimens in universal transport media will be archived for future respiratory pathogen testing.
  EDTA-whole blood, EDTA-derived plasma, sodium citrate-derived plasma, dried blood spots, serum, and blood culture broths will be archived for future etiologic or immunologic investigations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with sepsis

SUMMARY:
The aim of this study is to prospectively evaluate the barriers to care, evaluation, clinical practices, and outcomes for patients presenting with sepsis to hospitals in the Kilimanjaro Region of northern Tanzania. This will include an assessment of timing and selection of antimicrobials and administration and volume of intravenous fluids. The study also aims to characterize sepsis sub-types in the epidemiologic context of northern Tanzania using statistical clustering techniques of clinical variables and of host immune response patterns.

DETAILED DESCRIPTION:
A prospective observational cohort study of adolescent and adult patients with sepsis presenting to hospitals in the Kilimanjaro Region, Tanzania. Participants ≥10 years of age with suspected infection and the presence of two of the following will be enrolled: (1) tympanic temperature > 38°C or < 36°C, (2) heart rate > 90 beats/minute, (3) respiratory rate > 20 breaths/minute. Participants will be observed in the Emergency Department and during admission. The following data will be collected: demographics and medical history; history of present illness; laboratory and microbiological workup; antimicrobial selection and timing; intravenous fluid timing and volume. Vital status will be determined at 7 days, hospital discharge, and 28 days post-presentation. An enrollment of up to 1250 patients with sepsis is expected over a two-year period.

This study is expected to produce additional descriptive data of sepsis epidemiology and current practice in sSA. The data will yield important insights regarding key care practices for sepsis, including antimicrobial and intravenous fluid management. Outcomes of patients with sepsis will be described, including an assessment for correlations between current care practices and mortality.

Characterization of potential sepsis sub-types will be undertaken in two domains: 1) clinical characterization via a robust battery of routine clinical laboratories (chemistry, hematology, coagulation studies), vital signs, routine clinical signs and anthropometry; 2) host immune response characterization by analysis of mRNA transcriptome expression in RNA-stabilized whole blood samples. The goal of the sub-type characterization is to identity discrete and clinically relevant sepsis phenotypes, and in doing so eventually help optimize evaluation and management of sepsis specific to the populations and health systems in sub-Saharan Africa. Detailed etiologic investigations will also take place, including blood culture, blood parasite smears, and viral respiratory testing of nasopharyngeal samples; for patients living with HIV, additional evaluations will include serum cryptococcal antigen, urine lipoarabinomannan assay (TB-LAM) and MycoFLytic blood culture. Collectively, the data collected in this observational cohort study will contribute to further developing sepsis management bundles better suited to settings sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

Persons ≥ 10 years of age presenting to hospital suspected to have an infection and meeting two of the following vital signs criteria:

* tympanic >38°C or < 36°C
* a heart rate > 90 beats per minute
* a respiratory rate of > 20 breaths per minute

Exclusion Criteria:

* patient with a language barrier
* pregnant female
* a refugee
* a prisoner

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult patients with sepsis presenting to emergency department or outpatient department at hospitals in Kilimanjaro Region, northern Tanzania.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Sepsis sub-types derived from clinical characteristics. | Up to 4 years
  Number of sepsis subtypes identified by statistical clustering analysis of clinical characteristics.
Sepsis sub-types derived from host immune response to infection. | Up to 4 years
  Number of sepsis subtypes identified by statistical clustering analysis of patient immune response as measured by mRNA gene expression transcrimptomic signature.
Mortality due to sepsis | Within 28 days of presentation to hospital triage
  Time (measured in hours) to fatal event among patients with sepsis as measured by study staff observation or interview.
28-day mortality due to sepsis | Within 28 days of presentation to hospital triage
  Percentage of sepsis patients alive at 28 days after presentation to hospital triage as measured by study staff observation or interview.

SECONDARY OUTCOMES:
Delay in care-seeking for sepsis | Within 24 hours of presentation to hospital triage
  Percent of sepsis patients with a World Health Organization severity sign who delayed seeking medical care outside the home > 24 hours after onset of the severity sign as measured by patient/patient representative report.
Factors that slowed care-seeking | Within 24 hours of presentation to hospital triage
  Number of factors that slowed down the decision to seek care at hospital for present illness as measured by patient/patient representative report.
Time to antibiotics among patients with sepsis | Within 24 hours of presentation to hospital triage
  Time in hours from initial presentation at hospital triage to administration of antibiotics among patients with sepsis as measured by study staff observation and hospital records.
Intravenous venous fluid resuscitation among patients with sepsis | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients who receive intravenous fluids within 6 hours of presentation at hospital triage as measured by study staff observation and real-time review of hospital charting records.
Volume of intravenous fluid resuscitation among patients with sepsis | Within 6 hours of presentation to hospital triage
  Volume (measured in liters) of intravenous fluids received within 6 hours presentation at hospital triage as measured by study staff observation and real-time review of hospital charting records.
In-hospital mortality due to sepsis | Within 28 days of presentation to hospital triage
  Percentage of sepsis patients who survive to hospital discharge as measured by study staff observation.
7-day mortality due to sepsis | Within 7 days of presentation to hospital triage
  Percentage of sepsis patients alive at 7 days after presentation to hospital triage as measured by study staff observation or interview.
Clinical characteristic sub-type non-classification | Up to 4 years
  Percentage of sepsis patients who could not be classified into a sepsis sub-type derived by statistical clustering of clinical characteristics.
Immune response sub-types non-classification | Up to 4 years
  Percentage of sepsis patients who could not be classified into a sepsis sub-type derived by statistical clustering of patient immune response as measured by mRNA gene expression transcrimptomic signature.

OTHER OUTCOMES:
Sepsis due to respiratory syndrome | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a respiratory syndrome as measured by study staff standardized observation of signs and symptoms.
Sepsis due to neurologic syndrome | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a neurologic syndrome as measured by study staff standardized observation of signs and symptoms.
Sepsis due to genito-urinary syndrome | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a geninto-urinary syndrome as measured by study staff standardized observation of signs and symptoms.
Sepsis due to skin/soft tissue syndrome. | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a skin/soft tissue syndrome as measured by study staff standardized observation of signs and symptoms.
Sepsis due to gastrointestinal syndrome. | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a gastrointestinal syndrome as measured by study staff standardized observation of signs and symptoms.
Sepsis due to undifferentiated syndrome. | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with an undifferentiated syndrome as measured by study staff standardized observation of signs and symptoms.
HIV-infection among sepsis patients | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients who are infected with HIV as measured by World Health Organization approved rapid HIV antibody testing.
Sepsis severity of illness | Within 24 hours of presentation to hospital triage
  Percentage of sepsis patients presenting with a Universal Vital Assessment score > 4 as measured by study staff standardized observation of vital signs and measurement of HIV infection status.
Pre-specified sub-group analysis: enrolled participants with Sequential Organ Failure Assessment (SOFA) score of 2 or greater. | Up to 4 years
  The above outcomes will also be examined for this pre-specified sub-group of enrolled participants-- those who have a SOFA score of 2 or greater at the time of screening and enrollment.
Pre-specified sub-group analysis: enrolled participants with C-reactive protein measurement of 15 mg/L or higher | Up to 4 years
  The above outcomes will also be examined for this pre-specified sub-group of enrolled participants-- those who have a C-reactive protein serum measurement of above 15 mg/L (above the upper limit of a normal reference range in East Africa) at the time of screening and enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Rubach, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Centre, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level participant data will be de-identified and locator/identifying variables will be removed prior to sharing. Data availability will follow US National Institutes of Health guidelines for genomic data sharing, and it will include uploading annotated gene expression data files to the Gene Expression Omnibus system at the National Center for Biotechnology Information. Any sharing will also comply with regulations of the National Institute for Medical Research in Tanzania, including compliance with data transfer agreements between Kilimanjaro Christian Medical Centre and Duke University.
Supporting Information: Study Protocol
Time Frame: Gene expression data will become available at time of submission of the first manuscript that describes any such data. Additional data will be available per publisher or US National Institutes of Health policies or by written request to the Principal Investigators, provided that the sharing is compliant with the data sharing policies of the Tanzanian National Institute for Medical Research. Once available, there are no anticipated restrictions on the duration of availability.
Access Criteria: For data uploaded to the Gene Expression Omnibus, access will be designated per the policies of the US National Center for Biotechnology Information. For data uploaded in compliance with publishers, access will be designated per the policies of the publisher. Data can also be shared upon written request to the Principal Investigators and only shared once appropriate data sharing procedures have taken place in accordance with the policies of the Tanzanian National Institute for Medical Research.